CLINICAL TRIAL: NCT06235541
Title: A Phase I Study to Evaluate the Safety and Tolerability of GENA-104A16 (Anti-contactin4 [CNTN4] Monoclonal Antibody [mAb]) in Patients With Advanced Solid Tumors
Brief Title: A First-in-human Study of GENA-104A16 in Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Genome & Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [GNC] GENA104-101
Record Dates: First submitted 2024-01-15; First posted 2024-02-01 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GENA104 (Experimental): 80 patients in total with histologically/cytologically confirmed unresectable, recurrent, or metastatic advanced solid tumors, for who no standard therapy exists, or standard therapy has failed will be enrolled in this study.
  Interventions: Drug: GENA-104A16

INTERVENTIONS:
Drug: GENA-104A16 — GENA-104A16 is administered as a 1 hour (h) [-5 minutes and +60 minutes , i.e., 55-120 minutes as window time] as intravenous (IV) infusion on q2w.

SUMMARY:
This is a first in human phase I , open label study to evaluate the safety and tolerability of GENA 104A16 administered as a single agent by intravenous (IV) once every 2 weeks ( q2w (1 cycle = 2 weeks) in patients with advanced solid tumors, for who no standard therapy exists, or standard therapy has failed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically/cytologically confirmed unresectable, recurrent, or metastatic advanced solid tumors
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1
* Adequate organ function including hematological, hepatic, and renal functions.
* Negative childbearing potential
* Measurable disease as per RECIST v1.1 defined as at least 1 lesion
* Patients who are willing and able to comply with scheduled cycles, treatment plans, laboratory tests, and other procedures

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test prior to treatment
* Received prior systemic anti-cancer therapy within 4 weeks or 5 half-life periods (whichever is shorter) prior to the first dose of treatment
* Received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis
* Received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention
* Currently participating and receiving study treatments or has participated in a study of an investigational agent and received the study therapy or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Had an allogeneic tissue/solid organ transplant
* A diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* A known additional malignancy that is progressing or has required active treatment within the past 3 years
* A known active CNS metastases and/or carcinomatous meningitis
* A known prior severe hypersensitivity reactions to monoclonal antibodies or any component in their formulation (Grade ≥3)
* An active autoimmune disease that has required systemic treatment in past 2 years
* A history of (non infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* An active infection requiring systemic therapy, or has received a course of antibiotics within 4 weeks prior to the first dose of treatment
* A known history of human Immunodeficiency Virus (HIV) infection
* A known history of Hepatitis B or known active Hepatitis C virus (HCV) infection
* Diagnosed with Gliosis through a brain MRI and has experienced neurological conditions within 6 months before the first administration
* Has any one or more clinically significant cardiovascular disease
* A history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the patients participation for the full duration of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD and RP2D | 1 year
  Incidence of dose limiting toxicity (DLT).
Incidence of Adverse Events | 1 year
  Assessed as per CTCAE v5.0
Incidence of Laboratory abnormalities | 1 year
  Assessed as per CTCAE v5.0

SECONDARY OUTCOMES:
Cmax for Pharmacokinetic (PK) profile | 1 year
  Maximum serum concentration
Tmax for Pharmacokinetic (PK) profile | 1 year
  Time to reach the maximum concentration
AUC0-tlast for Pharmacokinetic (PK) profile | 1 year
  The area under the concentration-time curve from the time of dosing (time 0) to the time of the last observation
Half-life for Pharmacokinetic (PK) profile | 1 year
  Measurement of half-life as PK parameter
Clearance for Pharmacokinetic (PK) profile | 1 year
  Measurement of clearance as PK parameter
Potential immunogenicity | 1 year
  Levels of human anti-GENA-104A16 antibody
Objective response rate (ORR) | 1 year
  Assessed according to RECIST v1.1
Duration of response (DoR) | 1 year
  Assessed according to RECIST v1.1
Progression free Survival (PFS) | 1 year
  Assessed according to RECIST v1.1

OTHER OUTCOMES:
Tumor Biospecimens | 1 year
  Levels of biomarkers expression with the observed antitumor activity
Blood Biospecimens | 1 year
  Levels of biomarkers expression with the observed antitumor activity
Fecal Biospecimens | 1 year
  Levels of biomarkers expression with the observed antitumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Doyoun Oh, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No